CLINICAL TRIAL: NCT02290977
Title: Scheduled Interval Trans-catheter Arterial Chemo-embolization and Radiation Therapy for Hepatocellular Carcinoma Combined With Portal Vein Tumor Thrombosis: Prospective Phase II Trial
Brief Title: Transarterial Chemoembolization (TACE) With Radiation Therapy (RT) in Advanced Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Paik Yong Han, Associate Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-07-009
Record Dates: First submitted 2014-11-06; First posted 2014-11-14 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Hepatocellular Carcinoma; Portal Vein Tumor Thrombosis
Keywords: RT, TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Scheduled TACE-RT (Experimental): RT will be delivered at two weeks after TACE for HCC combined PVTT.
  Interventions: Radiation: Scheduled interval TACE - RT

INTERVENTIONS:
Radiation: Scheduled interval TACE - RT — RT will be administered at 2 weeks after TACE in HCC combined PVTT

SUMMARY:
The presence of portal vein tumor thrombosis (PVTT) in patients with hepatocellular carcinoma (HCC) is one of the most significant prognostic factors for poor prognosis, without treatment, their survival is less than 3 months. In the HCC patients who combined with PVTT, Radiation therapy (RT) showed 50% of local control and about 10 months survival duration. Despite the standard treatment of the HCC combined with PVTT is sorafenib, but Korean Liver Cancer Study Group (KLCSG) recommend RT as an alternative option in those patients. Investigators previously reported the retrospective study that the scheduled interval Trans-catheter Arterial Chemo-embolization (TACE) followed by RT for HCC combined with PVTT and 60% of the patients showed objective response without significant elevation of complication. However, the prospective outcomes of TACE followed by RT for HCC are scantly reported. Based on those background, we start this prospective study to evaluate the clinical outcomes and adverse event in the RT after TACE in the unresectable HCC patients who combined with PVTT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of HCC by at least one criterion listed below (korean liver cancer study group (KLCSG) guideline 2009) 1.1 Pathologically (histologically or cytologically) proven diagnosis of HCC 1.2 Liver nodule in high risk group 1.2.1 If alpha fetoprotein (AFP) ≥200 ng/mL , ≥ 1 typical HCC enhancing pattern on dynamic contrast enhanced CT or MRI 1.2.2 If AFP<200 ng/mL, ≥2 typical HCC enhancing pattern on dynamic contrast enhanced CT, MRI, and angiography 1.3 ≥ 2 cm nodule in liver cirrhosis (LC), ≥ 1 typical HCC enhancing pattern on dynamic contrast enhanced CT or MRI
2. Patients must have a diagnosis of PVTT 2.1 Early arterial enhancement and delayed washout on multiphasic CT or MRI
3. Eastern cooperative oncology group performance status 0 1 2
4. Age ≥ 20 and 70 or less
5. Unsuitable for resection or transplant or radiofrequency ablation (RFA)
6. Unsuitable for or refractory to TACE or drug eluting beads (DEB)
7. Agreement of study-specific informed consent
8. Assessment by radiation oncologist and medical oncologist or hepatologist within 28 days prior to study entry?
9. Child-Pugh score A-B within 7 days prior to study entry
10. Normal liver (Liver minus gross tumor volume) ≥ 700 cc
11. Blood work requirements

    * Absolute neutrophil count (ANC) ≥ 1,500 /mm3, Platelet ≥ 70,000/mm3, Hgb ≥ 8 g/dl
    * Liver function test (LFT): Total bilirubin<3.0 mg/dL, International normalized ratio(INR) < 1.7, Albumin ≥ 2.8g/dL, Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT)< 6 X normal
    * Serum creatinine < 1.5 X normal, or creatinine clearance ≥ 60 mL/min
12. Male, consent contraception at least 6 months
13. Childbearing potential woman, consent contraception at least 6 months
14. Life expectancy more than 12 weeks
15. Stable breathing more than 5 minutes

Exclusion Criteria:

* 1. Complete obstruction of main portal vein 2. Pregnant and/or breastfeeding woman 3. Previous upper abdominal RT history 4. Uncontrolled active co-morbidity 5. Another primary cancer history within 2 years 6. Uncontrolled ascites or hepatic encephalopathy 7. Connective tissue disease which known as radiation hypersensitivity 8. Uncontrolled moderate to severe gastroduodenal ulcer or esophagogastric varices

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-10 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate after scheduled TACE-RT for HCC with PVTT | One year after treatment
  Overall survival rate will be evaluated at 1 year after treatment.
Adverse event assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 after scheduled TACE-RT for HCC with PVTT | Three months after treatment
  Adverse event will be evaluated at 3 months after treatment.

SECONDARY OUTCOMES:
Radiologic response assessed by modified Response Evaluation Criteria for Solid Tumors (mRECIST) after scheduled TACE-RT for HCC with PVTT | Three months after treatment
  Radiologic response will be evaluated at 3 months after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea